CLINICAL TRIAL: NCT07279545
Title: The Effect of Placental Cord Drainage on the Third Stage of Labor and the Amount of Postpartum Bleeding
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Sinem Gültekin, Sp. Midwife, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GSBU-SBF-SG-01
Record Dates: First submitted 2025-11-14; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Postpartum Hemorrhage
Keywords: active management; third stage of labor; placental cord drainage; postpartum hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Masking Description: Two groups with a intervention and control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placental Cord Drainage Group (Experimental): In the intervention group, after the cord is cut, the clamp remaining at the maternal end will be released, allowing for controlled placental drainage into the kidney basin. This procedure will continue until signs of placental separation are observed. If at least one of these signs of separation is observed, the cord will be re-clamped. Signs of separation are expected to occur within 5 minutes, but if no signs of separation are observed within 5 minutes, the procedure will be terminated and the cord will be re-clamped. The midwife will remain with the patient at all times during this period.
  Interventions: Procedure: Placental cord drainage
- Control Group (No Intervention): In the women in the control group, the more routine practice in the clinic will be applied, that is, the umbilical cord will remain clamped until the placenta is delivered.

INTERVENTIONS:
Procedure: Placental cord drainage — Placental cord drainage is the process of clamping and cutting the umbilical cord after the birth of the baby, then opening the clamp at the maternal end of the cord and allowing the blood in the placenta to flow outward (Soltani et al, 2011; Vasconcelos et al, 2018; Pandey et al, 2019; Upadya et al, 2019; Chaudhary et al, 2020; Kazı et al, 2020; Mittal et al, 2020; Nabıl and Marzouk, 2020; Mansour et al, 2021; El Sayed et al, 2021; Karimi et al, 2022; Wedn and Hassanin, 2022).
  Arms: Placental Cord Drainage Group

SUMMARY:
The aim of the study was to evaluate the effect of controlled placental cord drainage by opening the clamp at the maternal end after the umbilical cord is cut during birth on the duration of the third stage of labor (departure of the placenta), the amount of blood loss in the third stage, the amount of bleeding in the 2nd hour postpartum, and the development of postpartum complications.

DETAILED DESCRIPTION:
Although the third stage is the shortest stage of labor, it is also the riskiest. Prolonging this stage increases the risk of complications, particularly postpartum hemorrhage. Therefore, the duration of the third stage of labor should be as short as possible. Internationally accepted labor management guidelines, such as WHO and ACOG, recommend that active management be adopted to shorten the third stage of labor to prevent postpartum hemorrhage. Placental cord drainage is also mentioned in the literature as a method used to accelerate the delivery of the placenta by actively managing the third stage of labor. This method involves clamping and cutting the umbilical cord after the birth of the baby, then opening the clamp at the maternal end of the cord and allowing the blood in the placenta to flow outward. It is suggested that this method will make the placenta smaller and more compact by reducing its volume, thus providing more effective contractions in the uterus and consequently, earlier separation and expulsion of the placenta with less blood loss. This method is implemented as national policy in 32% of maternity units in Belgium, 24% in Portugal, 15% in Norway and Spain, and approximately 14% in Ireland. In our country, physicians and midwives have also been observed using this method when signs of placental separation are delayed. To facilitate placental separation, they open the clamp at the maternal end and allow some blood to flow from the placenta.

A review of studies reveals conflicting results. A Cochrane review of three studies involving 1,257 women reported that placental cord drainage shortened the length of the third stage of labor by an average of three minutes and reduced blood loss by an average of 77 ml. A meta-analysis of nine randomized controlled trials confirmed the effectiveness of placental cord drainage in shortening the length of the third stage, but the results showed that it did not reduce blood loss. However, more recent studies have reached conflicting conclusions. While some studies have found that placental cord drainage produces a significant reduction in postpartum blood loss and the duration of the third stage of labor, others have reported that it has no effect in reducing postpartum blood loss and shortening the third stage of labor. In addition, in all studies conducted on the subject, the incidence of complications such as postpartum hemorrhage, placental retention, hand hallas, additional medication and blood transfusion requirement was found to be lower. However, further studies are needed to determine whether placental cord drainage is effective in shortening the duration of the third stage of labor and reducing postpartum hemorrhage. Therefore, this study aimed to evaluate the effect of placental cord drainage on the third stage of labor and the amount of postpartum hemorrhage.

The study's results are significant because they add to the growing body of evidence by offering a new perspective on a controversial topic. The interventions implemented in this study are expected to result in a quicker delivery of the placenta, less bleeding, and a lower risk of postpartum complications. All of these benefits will contribute to a smoother delivery process. Complications experienced during the third stage can lead to anemia, necessitate blood transfusions, and delay the initiation of breastfeeding, affecting the health of the newborn. Considering the impact of all these negative effects on hospital costs, the national economy, and health indicators, it would be meaningful to expand the use of placental cord drainage in clinics for the active management of the third stage of labor, provided its effectiveness is demonstrated. Furthermore, considering its minimal effort, low cost, and its potential as an alternative midwifery method in regions where access to oxytocin and methergine is not available, widespread adoption is significant.

Data Collection

When pregnant women are admitted to the delivery room, the purpose, importance, and procedures of the study will be explained to those who meet the inclusion criteria. Written consent will be obtained from pregnant women who agree to participate. Pregnant women will then be assigned to either the intervention or control group based on their corresponding values in a simple random number table generated through www.random.org.

All pregnant women will then be administered a "Pregnancy Information Form," and the labor process will be monitored using a "Labor Monitoring and Evaluation Form." The start and end times of each stage of labor will be recorded using a digital clock, and the duration will be calculated. The time of birth will be considered the start of the third stage.

As soon as the baby is born, the V-drope blood collection bag will be placed appropriately under the woman's hips by the auxiliary staff.

All women in the intervention and control groups will receive prophylactic treatment determined by the physician's order, in accordance with hospital protocols (20 units of synpitan IV bolus in 500cc 5% dextrose).

The umbilical cord will be clamped and cut within 1 minute after the baby's birth.

In the intervention group, after the cord is cut, the clamp will be released, allowing placental drainage into the kidney basin in a controlled manner. This procedure will continue until signs of placental separation are observed. The cord will be re-clamped when at least one of these signs of separation is observed. Signs of separation are expected to occur within 5 minutes, but if no signs of separation are observed within 5 minutes, the procedure will be terminated and the cord will be re-clamped. The midwife will remain with the patient during this time. The placental drainage blood collected in the kidney basin will be measured using a precision digital scale, and the tare value of the kidney basin will be recorded.

In the women in the control group, the routine procedure will be performed, meaning the umbilical cord will remain clamped until the placenta is delivered.

While waiting for signs of placental separation in the intervention and control groups, the woman's pulse and blood pressure will be measured and recorded by another midwife.

In the intervention and control groups, after signs of placental separation appear, the placenta will be delivered using controlled cord traction (Brandt-Andrew maneuver). The cotyledons and membranes will be examined, and the placental thickness and weight will be measured. Uterine tone and bladder fullness will be assessed.

In the intervention and control groups, the time of placental delivery will be recorded using a digital clock. The time between the birth of the baby and the delivery of the placenta will constitute the duration of the third stage of labor.

The amount of blood lost in stage 3 will be calculated by measuring the blood collected in the V-drop in the control group (ml). In the intervention group, the placental drainage blood collected in the kidney basin (grams) will be added to the blood collected in the V-drop (ml). The total amount of blood loss will be calculated in ml. The calculation of the blood in the kidney basin in ml will be made as follows: (The weight of the kidney basin filled with blood after taring ÷ 1.05).

If present, an episiotomy and repair of first- and second-degree lacerations will be performed. In cases where an episiotomy is necessary or first- or second-degree lacerations have occurred, blood from the episiotomy wounds or perineal lacerations will be tamponaded with a sponge and removed to avoid compromising the results.

After an episiotomy or laceration repair, the vaginal and perineal wound length will be measured and recorded with a disposable wound measuring ruler. A physician's order will then be administered according to hospital routines (1x2 amp IM methylerol (ergometrine) for all pregnant women whose blood pressure is not above 140-90 mm Hg). Women will then be dressed in absorbent, leak-proof underwear and taken to bed.

Women will remain under observation in the delivery room for the next two hours to monitor for any postpartum complications. After delivery, vital signs and uterine tone will be monitored according to hospital routine protocol.

Breastfeeding will be initiated within the first half hour after birth, and the start time and duration of breastfeeding will be recorded.

At the end of the second hour postpartum, the leak-proof underwear will be removed and weighed on a precision scale. The amount of blood lost at this stage will be calculated in ml as follows: (Weight of the leak-proof absorbent underwear used - weight before use) ÷ 1.05.

Hb and Hct results of women in the intervention and control groups at the 24th hour after birth will be recorded from the patient file.

The amount of bleeding during pregnancy, as well as all postpartum measurements and assessments, will be performed and recorded by an assistant midwife who is unaware of the pregnant woman's group. This is intended to increase the reliability of the data.

ELIGIBILITY:
Inclusion Criteria:

* No problem speaking and understanding Turkish
* Low-risk pregnant women
* Vertex presentation
* 37-41st weeks of gestation
* There are no complications in the mother or the baby that prevent normal birth.
* The VAS score for the pain felt by the pregnant woman at the time of admission to the study must be less than 3 (to show that the pregnant women were accepted into the study at a time when their pain was at its lowest and their decision-making ability was at a relatively good level)

Exclusion Criteria:

* History of postpartum hemorrhage
* History of postpartum hemorrhage in mother or sister
* Birth interval less than 2 years
* Anticoagulant use during pregnancy
* Smoking during pregnancy
* Those with low Hb values (Hb<11gr/dL)
* Hematocrit <30

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only female participants will be included in this study because the condition under investigation occurs exclusively in woman.
Enrollment: 80 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2026-06-20 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Determining the duration of the third stage of labor | The time between the birth of the newborn and the delivery of the placenta
  In the intervention and control groups, the time of placental delivery will be recorded using a digital clock. The time between the birth of the newborn and the delivery of the placenta will constitute the duration of the third stage of labor.
Determining the amount of blood lost in the 3rd stage | Until one of the signs of placental separation is seen, maximum 5 minutes
  In the control group, the blood collected in the V-drop (ml) will be measured and calculated. In the intervention group, the placental drainage blood collected in the kidney basin (grams) will be added to the blood collected in the V-drop (ml). The total amount of blood loss will be calculated in ml. The blood in the kidney basin will be calculated in ml as follows: (The weight of the kidney basin filled with blood after taring ÷ 1.05) (Asıcıoğlu et al, 2015).
Determination of the amount of hemorrhage at the 2nd hour postpartum | Postpartum 0-2 hours
  At the end of the second hour postpartum, the leak-proof underwear will be removed and weighed on a precision scale. The amount of blood lost at this stage will be calculated in ml as follows: (The weight of the leak-proof absorbent underwear used - the weight before use) ÷ 1.05. (Asıcıoglu et al, 2015).

SECONDARY OUTCOMES:
Hemoglobin and hematocrit levels at 24 hours postpartum, changes compared to prepartum | Admission to the delivery room - postpartum 24th hour
  Hb and Hct results of women in the intervention and control groups at the 24th hour after birth will be recorded from the patient file.
The possibility of developing complications in the third stages of labor | The time from the moment of placental cord drainage until placental separation
  Participants will be evaluated for complications such as hypotension, syncope, retained placenta, manual delivery of the placenta, and the need for additional medication.
The possibility of developing complications in the fourth stage of labor | Postpartum until the 24th hour after delivery of the placenta
  Participants will be evaluated for complications such as atony, abnormal uterine bleeding, and the need for additional medication.

CONTACTS AND LOCATIONS:
Overall Officials: Ferhat TÜFEKÇİ, Spc. Dr., Principal Investigator — Zonguldak Maternity and Child Diseases Hospital
Locations (1):
- Zonguldak Maternity and Child Diseases Hospital, Zonguldak, Zonguldak/Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.

REFERENCES:
- See also: Placental Cord Drainage Versus Clamping for Prevention of Blood Loss in the Third Stage of Labour — https://mjcu.journals.ekb.eg/article_105129_bc900209839722d80bca647b591fc076.pdf
- See also: Influence of placental cord drainage in management of the third stage of labor: a multicenter randomized controlled study — https://pubmed.ncbi.nlm.nih.gov/25111038/
- See also: Effect of Placental Cord Blood Drainage on Duration of Third Stage of Labour — https://pjmhsonline.com/index.php/pjmhs/article/view/1557/1542
- See also: Practice Bulletin No. 183: Postpartum Hemorrhage — https://pubmed.ncbi.nlm.nih.gov/28937571/
- See also: Placental cord drainage after vaginal delivery as part of the management of the third stage of labour — https://pubmed.ncbi.nlm.nih.gov/21901693/
- See also: Placental cord drainage in the third stage of labor: Randomized clinical trial — https://pubmed.ncbi.nlm.nih.gov/29718920/
- See also: The maternal side of placental cord blood drainage in the management of the third stage of labor: Relook the basic step in minimizing the maternal blood loss — https://www.gynaecologyjournal.com/articles/342/3-5-14-554.pdf
- See also: Role of Placental Cord Drainage in the Management of Third Stage of Labor after Normal Delivery — https://aimdrjournal.com/wp-content/uploads/2021/07/OG2_OA_Virendra-edit-1.pdf
- See also: Placental cord drainage during third stage of labour: a randomized control trial at a tertiary care centre — https://www.ijrcog.org/index.php/ijrcog/article/view/7904/5335
- See also: Comparison of Duration of Third Stage of Labour with and without Placental Cord Drainage (PCD) in Women Undergoing Normal Vaginal Delivery at Term — https://pjmhsonline.com/2021/feb/356.pdf
- See also: A comparative study of the effectiveness of placental blood drainage versus no placental blood drainage in active management of third stage of labor at a tertiary care hospital — https://www.ijrcog.org/index.php/ijrcog/article/view/9295
- See also: Placental Cord Drainage: Its Effect on Duration and Blood loss of Third Stage of Labor — https://ejhc.journals.ekb.eg/article_203222.html
- See also: Effects of placental cord drainage in the third stage of labour: A meta-analysis — https://www.nature.com/articles/s41598-017-07722-7
- See also: Comparison and the Duration of Third Stage of Labour with or without Cord Blood Drainage in Females Undergoing Normal Vaginal Delivery at Term — https://jsogp.net/index.php/jsogp/article/view/329
- See also: A study of placental blood drainage in third stage of labour to prevent postpartum haemorrhage: a randomized controlled study — https://www.ijrcog.org/index.php/ijrcog/article/view/10860
- See also: Placental cord drainage impact on third stage of labor: a randomized controlled trial — https://pubmed.ncbi.nlm.nih.gov/39098635/
- See also: Placental cord drainage and its outcomes at third stage of labor: a randomized controlled trial — https://bmcpregnancychildbirth.biomedcentral.com/articles/10.1186/s12884-022-04877-8
- See also: Drainage Of Placental Cord Blood In Dealing With The Third Stage Of Labor — https://www.pnrjournal.com/index.php/home/article/view/9018
- See also: Role of placental blood drainage as a part of active management of third stage of labour after spontaneous vaginal delivery — https://pubmed.ncbi.nlm.nih.gov/31853104/
- See also: Placental Drainage Versus No Placental Drainage After Vaginal Delivery in the Management of Third Stage of Labour: A Randomized Study — https://dergipark.org.tr/tr/pub/zktipb/issue/43374/457289
- See also: Placental cord drainage and the effect on the duration of third stage labour, a randomized controlled trial — https://pubmed.ncbi.nlm.nih.gov/19374293/
- See also: WHO recommendations for the prevention and treatment of postpartum haemorrhage — https://iris.who.int/server/api/core/bitstreams/36ea885b-7472-4b89-9605-81535f6a53c6/content
- See also: Influence of placental cord drainage in management of the third stage of labor: A Randomized controlled trial — https://www.noveltyjournals.com/upload/paper/Influence%20of%20placental%20cord%20drainage.pdf
- See also: Variations in policies for management of the third stage of labour and the immediate management of postpartum haemorrhage in Europe — https://pmc.ncbi.nlm.nih.gov/articles/PMC1974828/pdf/bjo0114-0845.pdf